CLINICAL TRIAL: NCT04388020
Title: Effects of Projected Peripheral Defocus on Ocular Biometrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eSpec Phase IIB
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Test Arm (Experimental)
  Interventions: Device: Tabletop prototype of eSpecs: Active projection of defocused image in the peripheral visual field; Device: Tabletop prototype of eSpecs: No Active projection of defocused image in the peripheral visual field

INTERVENTIONS:
Device: Tabletop prototype of eSpecs: Active projection of defocused image in the peripheral visual field — For the right/test eye, a defocused image is projected onto the peripheral retina while the subject views a distant, in-focus image
Device: Tabletop prototype of eSpecs: No Active projection of defocused image in the peripheral visual field — For the left/control eye, no image is projected onto the peripheral retina. The subject views a distant, in-focus image.

SUMMARY:
Acucela Inc. intends to develop a medical device to significantly halt or reverse myopic progression, which is a significant public health concern across the world, especially in Asian demographics. Acucela is working towards a spectacle-like device (eSPECs), which will have a clear zone for unimpeded central visual tasks and a periphery that provides defocus in order to alter retinal physiology leading to myopia regulation. This study will establish the changes seen during a proof-of-concept that projected defocus in the periphery will stimulate physiological changes similar to those in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent +2.00 to -4.00 diopters
* Refractive cylinder ≤ 0.75 diopters
* Visual acuity 20/20 -3 or better

Exclusion Criteria:

* Pregnant or lactating
* Active ocular infection
* History of dry eye, strabismus, or amblyopia
* Previous or planned ocular surgery
* Use of medication known to affect vision or accommodation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Axial length (AL) | 1 hour
  Change in AL from baseline in the test eye vs. control eye
Choroidal thickness (CT) | 1 hour
  Change in CT from baseline in the test eye vs. control eye

CONTACTS AND LOCATIONS:
Overall Officials: Arkady Selenow, OD, Principal Investigator — Manhattan Vision Associates
Locations (1):
- Manhattan Vision Associates/institute of Vision Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No